CLINICAL TRIAL: NCT00000571
Title: Trial of Inspiratory Muscle Rest and Exercise in Chronic Obstructive Lung Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: McGill University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: 209; R01HL034019 (NIH)
Record Dates: First submitted 1999-10-27; First posted 1999-10-28 (Estimated); Last update posted 2015-12-29 (Estimated); Status verified 2001-04

CONDITIONS: Lung Diseases; Lung Diseases, Obstructive; Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Lung Diseases; Lung Diseases, Obstructive; Pulmonary Disease, Chronic Obstructive | interventions — Ventilators, Negative-Pressure

INTERVENTIONS:
Device: ventilators, negative pressure

SUMMARY:
To test the effectiveness of ventilatory muscle rest (VMR) using home negative pressure ventilation (NPV) in improving exercise performance, alleviating dyspnea, and improving the quality of life in patients with severe chronic obstructive lung disease.

DETAILED DESCRIPTION:
BACKGROUND:

The potential importance of respiratory, chiefly inspiratory-muscle, fatigue had only recently been appreciated. If inspiratory muscles fail, so does ventilation and tissue respiration. There are theoretical reasons to postulate inspiratory muscle failure in chronic obstructive pulmonary disease, and suggestions that it may occur in an acute form with exacerbations and in a chronic form during 'stability'. There are two therapeutic strategies available for prevention and treatment of inspiratory muscle fatigue: training inspiratory muscles to increase their efficiency and resting fatigued muscles. The former should work if chronic fatigue is not present, and the latter should allow recovery from chronic fatigue, so the two approaches are not necessarily mutually exclusive. This proposal was originally designed to test the efficacy of each of these therapies alone and also in combination; however, given the experience of a pretrial period, these goals were scaled back. Since there was reason to believe that VMR may be more effective than IMT, the trial focused on VMR and sham VMR only.

Ventilatory muscle rest was applied using a negative pressure ventilation suit sealed at the patient's hips, arms, and neck. A widebore tube connected to a fitting in the suit above the grid on the chest and upper abdomen transmitted negative pressure to the chest wall from the pump, thereby inflating the lungs.

The evidence for chronic inspiratory muscle fatigue in patients with COLD resided largely in several relatively poorly controlled studies indicating that nocturnal artificial ventilation, which presumably rested the inspiratory muscles, produced improvement in daytime function and blood gases. The trial produced some badly needed data on both the occurrence of inspiratory muscle fatigue in COLD patients and its treatment with VMR.

DESIGN NARRATIVE:

Randomized, blinded. A total of 1,231 patients in the metropolitan Montreal area were screened. Of these, 348 were recruited to enter a four week stabilization period, and 184 were subsequently randomized to either active or sham negative pressure ventilation (NPV). A five day in-hospital period was used to train patients in ventilator use and obtain baseline measures of exercise capacity, lung function, respiratory symptoms, and quality of life. Randomization was stratified on the basis of whether or not the patient had been receiving oxygen at home. Home ventilation treatment took place during a following 12-week period. Respirator use was recorded from patient logs and from concealed meters installed in the units. Patients received four home visits by physiotherapists during the 12-week period and returned to the hospital for follow-up at four and twelve weeks post-discharge for reassessment. The principal outcome measure was the distance in meters walked in six minutes. Secondary outcome measures were cycle exercise endurance time, severity of dyspnea, quality of life, arterial blood gas tensions, and respiratory muscle strength.

ELIGIBILITY:
No eligibility criteria

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1986-02

CONTACTS AND LOCATIONS:
Overall Officials: Peter Macklem, Principal Investigator — McGill University

REFERENCES:
- [Background] Shapiro SH, Macklem PT, Gray-Donald K, Martin JG, Ernst PP, Wood-Dauphinee S, Hutchinson TA, Spitzer WO. A randomized clinical trial of negative pressure ventilation in severe chronic obstructive pulmonary disease: design and methods. J Clin Epidemiol. 1991;44(6):483-96. doi: 10.1016/0895-4356(91)90211-q. PMID 2037853